CLINICAL TRIAL: NCT04570046
Title: Retrospective Study on MR Imaging of ET and PD Patients Subjected With MRgFUS Thalamotomy
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Xin Lou, Chairman of Radiology Department, Chinese PLA General Hospital
Other Study IDs: MRgFUS-VIM-Retrospective-2020
Record Dates: First submitted 2020-09-13; First posted 2020-09-30 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Movement Disorders
Keywords: Essential tremor; Parkinson disease; MRgFUS; Magnetic resonance imaging
MeSH Terms: conditions — Movement Disorders; Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TD-PD patients undergoing MRgFUS thalamotomy: A total of 10 patients with tremor dominant PD underwent MRgFUS thalamotomy. Their clinical and imaging data were collected.
- MR-ET patients undergoing MRgFUS thalamotomy: A total of 58 patients with medication-resistant ET underwent MRgFUS thalamotomy. Their clinical and imaging data were collected.

SUMMARY:
The technological advance of magnetic resonance-guided focused ultrasound (MRgFUS) has once again brought lesion therapy back to the clinical frontline for the treatment of movement disorder. Thus far, the safety of MRgFUS has been widely proven and has just been made available in China in late 2020. We attempted to analyze the neuroplasticity characteristics and altered neural circuit activity in patients subjected with MRgFUS thalamotomy via post-hoc retrospective analysis of archived MR imaging in our site, and to explore potential biomarkers that could be used to predict the treatment outcome.

DETAILED DESCRIPTION:
Essential tremor (ET) and Parkinson disease (PD) are the most prevalent tremor disorders. ET, considered as a pure tremor disease, is characterized by upper limb intention or postural tremor, while PD is characterized by a variety of motor and nonmotor symptoms, among them rest tremor. Tremor suppression can be achieved by lesioning or stimulating a relay nucleus of the thalamus, known as the ventral intermediate nucleus (VIM). One emerging and promising approach to lesion VIM is magnetic resonance-guided focused ultrasound (MRgFUS). This technique allows delivery of spherical phased converging beams to a specific brain target using MR imaging (MRI) for guidance. A number of studies have demonstrated the effectiveness and safety of ExAblate MRgFUS thalamotomy for medication-refractory tremor in patients with ET/PD. MRgFUS thalamotomy has been approved by US FDA for ET/PD patients in 2017 and 2021 respectively.

Several Phase IV trials of MRgFUS thalamotomy for ET/PD was successively posted around 2017 in Asia. Among them, the prospective, multi-site, single-arm clinical trial of ET patients got registered in clinicaltrials.gov with NCT03253991 including our team in Chinese PLA General Hospital as one site (Prof. Pan Longsheng as the Principal Investigator). Our study was approved and started in November 2018 with patient recruitment via outpatient clinics and the Internet, and the main content of the study was completed in early 2020. Finally, MRgFUS thalamotomy was approved for ET treatment in late 2020.

These studies have left many valuable research materials with significant research value, including multimodal magnetic resonance imaging. The analysis of these imaging data may help us to further understand the neuroplasticity characteristics of patients around treatment and the altered brain network dynamics. It would also further help us grasp the advantages and disadvantages of such brain lesion therapy techniques and serves guidance for the next clinical studies. Therefore, we registered this new NCT04570046 for our current retrospective study.

Summary of retrospective data：

- Medication-refractory ET and PD Patients subjected with MRgFUS thalamotomy were collected, including baseline info, ultrasound parameters (energy, power, duration time, temperature, target location), clinical assessment (clinical rating scale for tremor (CRST), clinical variables and measurements at hospitalization, Unified Parkinson Disease Rating Scale (UPDRS), associated adverse effects and so on), MR imaging data at multiple timepoints (T2; T2 Flair; DWI; ESWAN; MRS; 3D ASL 2.0s; 3D-T1; DTI; rs-functional MRI at baseline, postoperative 1-day, postoperative 1-week, postoperative 1-month, postoperative 3-months, postoperative 6-months). Some patients may lost images at some timepoints, while Some patients may have extra images at other timepoints (postoperative 9-months or 1-year).

ELIGIBILITY:
All the data of ET/PD patients subject with MRgFUS thalamotomy were collected from 2017-2020 early in Chinese PLA General Hospital.

The inclusion and exclusion criteria for each patient at the time of previous surgery were:

* Inclusion Criteria:

  1. Men and women age 22 years or older;
  2. A diagnosis of ET and PD as confirmed from clinical history and examination by a neurologist or neurosurgeon specialized in movement disorder;
  3. Intolerance to side effects of medication or poor response to medication, severe and disabling tremor;
  4. Regarding PD patients, the ratio of mean Unified Parkinson Disease Rating Scale (UPDRS) tremor scores to the mean UPDRS postural instability/gait disorder scores equal or greater than 1.5;
  5. Able to communicate sensations during the ExAblate TcMRgFUS treatment;
  6. All MRI examination performed according to study protocol;
  7. Having complete medical history and clinical follow up;
  8. Imaging data can be processed.
* Exclusion Criteria:

  1. Subjects with unstable cardiac status;
  2. Severe hypertension (diastolic BP > 100 on medication);
  3. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc;
  4. Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease;
  5. Patient with severely impaired renal function;
  6. History of abnormal bleeding and/or coagulopathy;
  7. History of immunocompromise including those who are HIV positive;
  8. History of intracranial hemorrhage;
  9. Cerebrovascular disease (multiple CVA or CVA within 6 months);
  10. Subjects with uncontrolled symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, papilledema);
  11. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time);
  12. Significant claustrophobia that cannot be managed with mild medication;
  13. Presence of any other neurodegenerative disease such as Parkinson-plus syndromes suspected on neurological examination;
  14. Presence of significant cognitive impairment;
  15. Subjects with life-threatening systemic disease;
  16. Subjects with a history of seizures within the past year;
  17. Subjects with presence or history of psychosis.

Ages: 22 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ET and PD patients subject with MRgFUS thalamotomy
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Tremor symptoms in ET/PD patients subject with MRgFUS thalamotomy. | 2 years
  The change in the hand tremor score derived by summing the CRST ratings that evaluate hand tremor. Comparison will be performed from examinations at baseline and postoperative timepoints. According to the change of tremor performance after surgery, patients can be considered to be divided into whether there is effective tremor relieve or tremor recurrence.
Multimodal imaging spectrum features in ET/PD patients subject with MRgFUS thalamotomy. | 2 years
  From T2, T2 Flair, DWI, ESWAN, 3D-T1; ESWAN and MRS manifests were mapped and numeralized in the brain atlas, and then were used to construct multiple-dimensional spectrum features of brain alterations after MRgFUS thalamotomy, including brain functional activity, brain structural connectivity, cerebral blood flow, and so on.
Clinical variables spectrum features linking to the tremor symptoms and imaging spectrum features. | 2 years
  Medical records and test data of patients during hospitalization, including demographic characteristics, common comorbidity, hematological analysis, coagulation function, lipids profile, blood biochemistry, were used to construct clinical variables spectrum features. The distribution characteristics of postoperative tremor symptoms and imaging spectrum features were compared with the multi-dimensional matrix.

SECONDARY OUTCOMES:
Adverse events in ET/PD patients subject with MRgFUS thalamotomy. | 2 years
  Adverse Events will be evaluated using Significant Clinical Complications for movement disorders subjects. Adverse Events will be reported and categorized by investigators as definitely, probably, possibly, or unrelated to the device or procedure and categorized by treatment group / treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Lou, MD/PhD, Principal Investigator — Chinese PLA General Hospital; LongSheng Pan, MD/PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang D, Xiong Y, Lu H, Duan C, Huang J, Li Y, Bian X, Zhang D, Zhou J, Pan L, Lou X. Predicting tremor improvement after MRgFUS thalamotomy in essential tremor from preoperative spontaneous brain activity: A machine learning approach. Sci Bull (Beijing). 2024 Oct 15;69(19):3098-3105. doi: 10.1016/j.scib.2024.05.049. Epub 2024 Aug 16. PMID 39191568
- [Derived] Wang X, Wang S, Lin J, Zhang D, Lu H, Xiong Y, Deng L, Zhang D, Bian X, Zhou J, Pan L, Lou X. Gray matter alterations in tremor-dominant Parkinson's disease after MRgFUS thalamotomy are correlated with tremor improvement: a pilot study. Quant Imaging Med Surg. 2023 Jul 1;13(7):4415-4428. doi: 10.21037/qims-22-1403. Epub 2023 May 4. PMID 37456281